CLINICAL TRIAL: NCT00939783
Title: An Open Label Extension To The B1451027 Protocol To Evaluate The Long Term Safety And Tolerability Of Dimebon (PF 01913539) In Patients With Alzheimer's Disease
Brief Title: An Extension To The B1451027 Protocol To Evaluate The Long Term Safety And Tolerability Of Dimebon In Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1451029
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dimebon 20 mg TID (Experimental): 10 mg TID for Week 1, followed by 20 mg TID for remainder of study
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — Tablet for oral administration
  Other Names: PF-01913539

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of Dimebon in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
This study was terminated on May 7, 2010 as part of modification of the dimebon development plan following lack of demonstration of efficacy in the completed DIM14 (CONNECTION) Study. The study was not terminated due to any safety findings. Dimebon has been well -tolerated in clinical trials. Demonstration of efficacy for dimebon in Alzheimer's disease is pending completion of the ongoing DIM18 (CONCERT) Study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of previous Phase 3 Dimebon study (B1451027).

Exclusion Criteria:

* Have any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (80):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Northport, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Pueblo, Colorado
  - Pfizer Investigational Site, Hockessin, Delaware
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Fort Walton Beach, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Plant City, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Burr Ridge, Illinois
  - Pfizer Investigational Site, Elk Grove Village, Illinois
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Greenfield, Indiana
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Hyannis, Massachusetts
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Great Falls, Montana
  - Pfizer Investigational Site, Eatontown, New Jersey
  - Pfizer Investigational Site, Oakhurst, New Jersey
  - Pfizer Investigational Site, Toms River, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Grove City, Pennsylvania
  - Pfizer Investigational Site, Indiana, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Scotland, Pennsylvania
  - Pfizer Investigational Site, Upper Saint Clair, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Murrells Inlet, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Carrollton, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Grand Prairie, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Williamsburg, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Charleston, West Virginia
  - Pfizer Investigational Site, La Crosse, Wisconsin
- Canada (16):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Medicine Hat, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Pfizer Investigational Site, Kentville, Nova Scotia
  - Pfizer Investigational Site, Pictou, Nova Scotia
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, L'Ancienne-Lorette, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint-Jean-sur-Richelieu, Quebec
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Puerto Rico (3):
  - Pfizer Investigational Site, Cayey
  - Pfizer Investigational Site, Cidra
  - Pfizer Investigational Site, San Juan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451029&StudyName=An%20Extension%20To%20The%20B1451027%20Protocol%20To%20Evaluate%20The%20Long%20Term%20Safety%20And%20Tolerability%20Of%20Dimebon%20In%20Patients%20With%20Alzheimer%27s%20Dise

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimebon: Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by 20 mg tablet orally three times a day. Treatment was administered until participant withdrawal or study termination.
Period: Overall Study
Arm/Group | Dimebon
Started | 649
Treated | 648
Completed | 0
Not Completed | 649
Not completed — Death | 6
Not completed — Adverse Event | 39
Not completed — Study Terminated by Sponsor | 498
Not completed — Withdrawal by Subject | 78
Not completed — Other | 16
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 3
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dimebon
Number analyzed (Participants) | 648
Age, Customized [Number; unit: Participants]
  50 to 59 years | 32
  60 to 69 years | 100
  70 to 79 years | 269
  80 to 85 years | 187
  Greater than 85 years | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342
  Male | 306

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 65 (end of treatment)
Population: Safety analysis set included all the participants who received at least one dose of study medication, including partial doses.
Measure: Number; unit: Percentage of participants
Arm/Group | Dimebon
Number analyzed (Participants) | 648
Percentage of participants | 73.1

2. Secondary Outcome: Percentage of Participants With Abnormal Clinically Significant Vital Signs
Description: Abnormal clinically significant vital signs included absolute systolic blood pressure (BP) values less than (<) 90 millimeter of mercury (mmHg), maximum increase or decrease of greater than or equal to (>=) 30 mmHg from baseline for systolic BP; absolute diastolic BP <50 mmHg with maximum increase or decrease of >=20 mmHg from baseline and absolute heart rate values <40 beats per minute (bpm), >120 bpm for supine or sitting measurement, >140 bpm for standing measurement.
Time Frame: Baseline up to Week 65 (end of treatment)
Population: Safety analysis set included all the participants who received at least one dose of study medication, including partial doses. Here 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure and 'n' is signifying those participants who were evaluable for a particular category.
Measure: Number; unit: Percentage of participants
Arm/Group | Dimebon
Number analyzed (Participants) | 646
Percentage of participants
  Systolic BP (<90 mmHg) (n=646) | 1.1
  Increase in systolic BP (>=30 mmHg) (n=642) | 11.5
  Decrease in systolic BP (>=30 mmHg) (n=642) | 12.0
  Diastolic BP (<50 mmHg) (n=646) | 2.0
  Increase in diastolic BP (>=20 mmHg) (n=642) | 8.1
  Decrease in diastolic BP (>=20 mmHg) (n=642) | 9.7
  Heart rate (<40 bpm) (n=646) | 0.0
  Heart rate (>120/>140 bpm) (n=646) | 0.0

3. Secondary Outcome: Percentage of Participants With Abnormal Clinically Significant Laboratory Values
Description: For hematology, liver function, renal function, electrolytes, clinical chemistry, abnormality was reported if observed value was more than or less than X times upper limit of normal (ULN) or lower limit of normal (LLN); X=specified in categories of each parameter in measured values section. For urinalysis abnormality was reported if result was >=1 in qualitative test of all parameters except red and white blood cells which were reported if result was >=6, indicating levels in urine were abnormal. Urine pH abnormality reported if >8 and urine specific gravity abnormality if <1.003 or >1.030.
Time Frame: Baseline up to Week 65 (end of treatment)
Population: Safety analysis set included all the participants who received at least one dose of study medication, including partial doses. Here 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure and 'n' is signifying those participants who were evaluable for a particular laboratory parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Dimebon
Number analyzed (Participants) | 646
Percentage of participants
  Hemoglobin (<0.8*LLN) (n=646) | 0.3
  Red blood cell count (< 0.8*LLN) (n=646) | 0.5
  Mean corpuscular volume (<0.9*LLN) (n=646) | 0.8
  Mean corpuscular volume (>1.1*ULN) (n=646) | 0.2
  Platelets (>1.75*ULN) (n=646) | 0.2
  White blood cell count (<0.6*LLN) (n=646) | 0.2
  White blood cell count (>1.5*ULN) (n=646) | 0.2
  Lymphocytes (<0.8*LLN) (n=646) | 1.4
  Lymphocytes (>1.2*ULN) (n=646) | 2.6
  Total neutrophils (<0.8*LLN) (n=646) | 0.6
  Total neutrophils (>1.2*ULN) (n=646) | 4.3
  Eosinophils (>1.2*ULN) (n=646) | 1.4
  Monocytes (>1.2*ULN) (n=646) | 1.5
  Total bilirubin(>1.5*ULN) (n=646) | 0.3
  Aspartate aminotransferase (>3.0*ULN) (n=645) | 0.5
  Alanine aminotransferase (>3.0*ULN) (n=645) | 0.9
  Alkaline phosphatase (>3.0*ULN) (n=646) | 0.2
  Albumin (>1.2*ULN) (n=646) | 0.2
  Blood urea nitrogen (>1.3*ULN) (n=646) | 1.4
  Creatinine (>1.3*ULN) (n=646) | 1.4
  Sodium (<0.95*LLN) (n=646) | 0.3
  Sodium (>1.05*ULN) (n=646) | 0.9
  Potassium (<0.9*LLN) (n=645) | 0.6
  Potassium (>1.1*ULN) (n=645) | 0.5
  Calcium (>1.1*ULN) (n=646) | 0.3
  Magnesium (<0.9*LLN) (n=646) | 0.5
  Magnesium (>1.1*ULN) (n=646) | 22.0
  Phosphate (<0.8*LLN) (n=646) | 0.2
  Phosphate (>1.2*ULN) (n=646) | 0.2
  Bicarbonate (<0.9*LLN) (n=646) | 0.8
  Bicarbonate (>1.1*ULN) (n=646) | 0.2
  Glucose (>1.5*ULN) (n=646) | 17.6
  Creatine kinase (>2.0*ULN) (n=646) | 2.5
  Urine specific gravity (>1.030) (n=643) | 3.4
  Urine pH (>8) (n=643) | 0.3
  Urine glucose (>=1) (n=643) | 5.3
  Urine ketones (>=1) (n=643) | 2.2
  Urine protein (>=1) (n=643) | 3.3
  Urine blood (>=1) (n=643) | 52.1
  Urine leukocyte esterase (>=1) (n=643) | 29.4
  Urine RBC (>=6) (n=518) | 18.1
  Urine WBC (>=6) (n=562) | 34.3

4. Secondary Outcome: Percentage of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Abnormal ECG findings included maximum value of >=300 millisecond (msec), maximum increase of >=25% for baseline value of >200 msec and maximum increase of >=50% for baseline value of <=200 msec for PR interval (int); maximum increase of >=25% for baseline value of >100 msec and maximum increase of >=50% for baseline value of <=100 msec for QRS interval; maximum value of >450 to <=480, >480 to <=500 and >500 msec, increase of >30 to <=60 and >60 msec for QT interval corrected using Fridericia's formula (QTcF).
Time Frame: Baseline up to Week 65 (end of treatment)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Dimebon
Number analyzed (Participants) | 646
Percentage of participants
  PR int (>=300 msec) (n=608) | 0.3
  Increase in PR int (>=25/50%) (n=605) | 0.3
  Increase in QRS int (>=25/50%) (n=646) | 1.4
  QTcF int (>450 to <=480 msec) (n=646) | 18.3
  QTcF int (>480 to <=500 msec) (n=646) | 1.9
  QTcF int (>500 msec) (n=646) | 0.3
  Increase in QTcF int (>30 to <=60 msec) (n=646) | 8.0
  Increase in QTcF int (>60 msec) (n=646) | 0.3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dimebon
Serious Adverse Events (participants affected / at risk) | 76/648
Other Adverse Events (participants affected / at risk) | 313/648
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=648)
Angina pectoris (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Sick sinus syndrome (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Pancreatic mass (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 6
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Clostridial infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 6
Facial bones fractures (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 3
Fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 6
Joint dislocation (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Uterine rupture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dementia Alzheimer's type (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Acute psychosis (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 3
Psychotic disorder (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Calculus prostatic (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemodynamic instability (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=648)
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 28
Oedema peripheral (General disorders) | 22
Bronchitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 73
Contusion (Injury, poisoning and procedural complications) | 22
Fall (Injury, poisoning and procedural complications) | 59
Weight increased (Investigations) | 13
Anthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 15
Dizziness (Nervous system disorders) | 20
Headache (Nervous system disorders) | 25
Memory impairment (Nervous system disorders) | 15
Somnolence (Nervous system disorders) | 43
Agitation (Psychiatric disorders) | 20
Anxiety (Psychiatric disorders) | 19
Confusional state (Psychiatric disorders) | 23
Depression (Psychiatric disorders) | 18
Insomnia (Psychiatric disorders) | 15
Hypertension (Vascular disorders) | 18

LIMITATIONS AND CAVEATS:
This safety study did not specify primary or secondary outcome measures. Relevant summaries of all safety assessments are thus provided. Urine blood abnormalities seen are deemed due to interference with dipstick test by a metabolite of dimebon.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.